CLINICAL TRIAL: NCT02545699
Title: Prospective Randomized Trial to Compare the Adenoma Detection Rate of G-EYE™ Colonoscopy With Standard Colonoscopy
Brief Title: Prospective Trial to Compare ADR of G-EYE™ Colonoscopy With Standard Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: G-EYE 15507
Record Dates: First submitted 2015-08-31; First posted 2015-09-10 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Adenoma; Polyps; Colorectal Cancer
Keywords: Adenoma; Polyp; CRC; Colonoscopy; Detection Yield
MeSH Terms: conditions — Adenoma; Polyps; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-EYE™ Colonoscopy (Experimental): G-EYE™ Colonoscopy
  Interventions: Device: G-EYE™ Colonoscopy
- Standard Colonoscopy (Active Comparator): Standard Colonoscopy
  Interventions: Device: Standard Colonoscopy

INTERVENTIONS:
Device: G-EYE™ Colonoscopy — G-EYE™ Colonoscopy
  Arms: G-EYE™ Colonoscopy
Device: Standard Colonoscopy — Standard Colonoscopy
  Arms: Standard Colonoscopy

SUMMARY:
The purpose of this study is to compare the adenoma detection rate (ADR) of the G-EYE™ colonoscopy with that of standard colonoscopy.

DETAILED DESCRIPTION:
This is a single-center, two-arm , randomized, open-label study intended to compare the detection rate obtained by performing G-EYE™ colonoscopy vs. the detection rate obtained by performing standard colonoscopy.

The study will enroll 350 subjects. Consecutive adult subjects who were referred for elective colonoscopy will be asked to enroll in this randomized clinical study if the candidate meets the study inclusion and exclusion criteria.

Subjects will sign an informed consent form and undergo randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 50 years old
2. Referred to colonoscopy for screening, following positive FOBT testing, change of bowel habits, for diagnostic evaluation or for surveillance colonoscopy (history of adenoma resection).
3. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease;
2. Subjects with a personal history of polyposis syndrome;
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
4. Subjects with diverticulitis or toxic megacolon;
5. Subjects with a history of radiation therapy to abdomen or pelvis;
6. Pregnant or lactating female subjects;
7. Subjects who are currently enrolled in another clinical investigation.
8. Subjects with current oral or parenteral use of anticoagulants that have not stopped using anticoagulants as required by the guidelines of the medical center;
9. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
10. Any patient condition deemed too risky for the study by the investigator
11. Previous colonic surgery (except for appendectomy)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
G-EYE™ Colonoscopy detection rate of adenomas and serrated lesions compared to the standard colonoscopy detection rate of the same | Approximately following 14 days (histology results)

SECONDARY OUTCOMES:
Polyp and adenoma detection | Up to 14 days (Histology results)
  The secondary outcome is a composite- each of the measured parameters will be reported as a single value for each arm.
Procedure times | At time of procedure
Safety (number of patients with adverse events) | 48-72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tova Rainis, Dr., Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Hospital, Haifa, Israel